CLINICAL TRIAL: NCT05978544
Title: A Phase 1 Study to Evaluate the Safety, Tolerability and Preliminary Clinical Activity of Itolizumab in Subjects With Acute Respiratory Distress Syndrome Caused by Infectious Pneumonia
Brief Title: Safety and Preliminary Clinical Activity of Itolizumab in ARDS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Biotech Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BPL-ITO-ARDS-1001
Record Dates: First submitted 2023-07-20; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — itolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Itolizumab Dose Level 1 (Experimental): Itolizumab of 50 mg administered by intravenous infusion for once, investigator discretion to continue with the same dose every 3 days up to 7 days.
  Interventions: Drug: Itolizumab
- Itolizumab Dose Level 2 (Experimental): Itolizumab of 100 mg administered by intravenous infusion for once, investigator discretion to continue with the same dose every 3 days up to 7 days.
  Interventions: Drug: Itolizumab
- Itolizumab Dose Level 3 (Experimental): Itolizumab of 150 mg administered by intravenous infusion for once, investigator discretion to continue with the same dose every 3 days up to 7 days.
  Interventions: Drug: Itolizumab

INTERVENTIONS:
Drug: Itolizumab — Patients to be treated with Itolizumab.
  Other Names: T1h

SUMMARY:
To evaluate the safety, tolerability, PK, PD, and clinical activity of Itolizumab in subjects with acute respiratory distress syndrome (ARDS) caused by Infectious Pneumonia.

DETAILED DESCRIPTION:
The study will enroll approximately 38 subjects in two parts:

Part 1 is an open label 3+3 single dose escalation phase. 9-24 patients with ARDS caused by infectious pneumonia across 3 dose cohorts.

Part 2 is a randomized phase and will enroll approximately 14 additional participants, randomized in a 1:1 ratio to one of the 2 doses based on efficacy data obtained from Part 1.

All participants in this study will receive Itolizumab intravenously for once, investigator discretion to continue with the same dose every 3 days up to 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject aged 18-75 years old (inclusive)
2. Clinical diagnosis with infectious pneumonia as determined by the investigator
3. Subject who havd received anti-infective treatment according to clinical practice.
4. Diagnosis with ARDS according to the following criteria: (i) Bilateral opacities-not fully explained by effusions, lobar/lung collapse, or nodules; (ii) respiratory failure not fully explained by cardiac failure or fluid overload; (iii) Oxygenation (PaO2/FiO2) ≤300.
5. ARDS diagnosed within 48 hours before administration, and fullfil the criteria of ARDS before administration
6. Fullfill at least 2 of the following 4 criteria: ① elevated hs-CRP (>6 ULN); ② elevated IL-6 (>3 ULN); ③ high serum ferritin (>500µg/L at any one time or more than 2-fold increase within 48 hours of onset); ④ high D-dimer (>3 ULN).
7. Negative result of serum HCG within 72 hours before enrollment for female with potential fertility
8. Participant or his/her legal representive (when the participant is not capable of giving consent) is able to understand and comply with the planned procedure as required by the protocol, and sign a written informed consent form (ICF)

Exclusion Criteria:

1. ARDS caused by non-infectious pneumonia (e.g., burns, drowning, poisoning, etc.)
2. Subject who has cardiogenic pulmonary edema, and it is the main cause of respiratory failure
3. Subject who is at high risk of death within 24 hours regardless of the treatment measures given as determined by the investigator
4. Subject who is receiving extracorporeal membrane pulmonary oxygenation (ECMO) therapy at the time of screening.
5. Subject who had received mechanical ventilation for more than 72 hours prior to administration.
6. Subject with active tumors (other than carcinoma in situ or basal cell carcinoma) that requiring treatment.
7. Any of the following chronic organ damage or immunosuppression:

   1. Cardiac: cardiac arrest within 7 days prior to screening; New York Heart Association cardiac function class IV at screening;
   2. Pulmonary: oxygen therapy or ventilator-dependent therapy for more than 1 month cumulatively within 6 months prior to screening; pulmonary embolism within 4 weeks prior to screening; pulmonary hypertension, end-stage lung disease, or interstitial lung disease requiring glucocorticoid therapy at screening;
   3. Renal: serum creatinine > 1.5 ULN or creatinine clearance < 30 mL/min at screening (Cockcroft-Gault formula, see study protocol annex 5 for details) or on long-term dialysis treatment;
   4. Liver: liver function classification of Child-Pugh grade C at screening;
   5. Immunosuppression status: with lymphoma, leukemia or acquired immunodeficiency; having received antitumor chemotherapy in the last 3 months, or being treated with immunosuppression for organ transplantation or immune disorders; having had allogeneic bone marrow transplantation or allogeneic hematopoietic stem cell transplantation.
8. Subject who had vaccination within 28 days prior to administration, or plan to get the vaccine during the study period
9. Any of the following abnormalities at screening

   1. Hepatitis B-related tests: ① positive for hepatitis B surface antigen (HBsAg); ② positive for hepatitis B core antibody (HBcAb); ③ positive for hepatitis B surface antibody (HBsAb) and no history of hepatitis B vaccination; ④ positive for hepatitis B e antigen or hepatitis B e antibody;
   2. Positive hepatitis C virus antibody (HCV-Ab);
   3. Positive acquired immunodeficiency syndrome antibody (HIV-Ab).
10. Subject who has a medical history of tuberculosis or those who deny a history of tuberculosis but has a positive gamma-interferon release test at screening.
11. Absolute lymphocyte count < 0.2×109/L at screening
12. Suspected allergic to the investigational drug or any of its excipients
13. Currently pregnant, breastfeeding,or planning to become pregnant or not using reliable method to avoid pregnancy during study and within 3 months after the last study treatment
14. Subject who had participated in other clinical studies (other than those not receiving interventions, such as observational study or questionnaires survey) within 3 months prior to screening, or who are participating in other experimental treatments.
15. As determined by the investigator, any medical, psychiatric, or other condition or circumstance that is likely to negatively affect the reliability of the study data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-12-31 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events | Study Day 58
  Number of subjects with treatment-related adverse events as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) V5.0

SECONDARY OUTCOMES:
Maximum serum concentration of Itolizumab, Cmax | Study Day 30
  Maximum serum concentration of Itolizumab
Minimum serum concentration of Itolizumab, Cmin | Study Day 30
  Minimum serum concentration of Itolizumab
Time to maximum serum concentration of Itolizumab, Tmax | Study Day 30
  Time to maximum serum concentration of Itolizumab
Total Itolizumab exposure across time, AUC0-t | Study Day 30
  Total Itolizumab exposure across time
Half life of Itolizumab, t1/2 | Study Day 30
  Half life of Itolizumab
Inflammatory Markers,IL-6 | Study Day 30
  IL-6
Inflammatory Markers,TNF-α | Study Day 30
  TNF-α
Inflammatory Markers, hs-CRP | Study Day 30
  hs-CRP
Inflammatory Markers,Serum ferritin | Study Day 30
  Serum ferritin
Inflammatory Markers,D-dimer | Study Day 30
  D-dimer
CD6 receptor expression levels | Study Day 30
  Mean change of CD6 receptor expression levels in relative to baseline
T cell subsets | Study Day 30
  Mean change of different T cell subsets in relative to baseline
The proportion of patients with stable or improved Lung Function | Study Day 30
  Defined as patients with stable or improved PaO2 without increasing FiO2 in relative to baseline
Mean change from baseline in Murray Score | Study Day 30
  Mean change of Murray Score in relative to baseline，The higher score means the worse outcome
Mean change from baseline in SOFA score | Study Day 30
  Mean change of SOFA（Sequential Organ Failure Assessment） score in relative to baseline，The higher score means the worse outcome
Mechanical ventilation-free days | Study Day 30
  Duration of non-Mechanical ventilation
Oxygen therapy-free days | Study Day 30
  Duration of non-Oxygen therapy
Duration of ICU stay | Study Day 30
  ICU stay days
Mortality rate | Study Day 15, 30
  Defined as the proportion of patients who met fatal outcome event by Day 15 and 30
Clinical status assessed using a 7-category ordinal scale | Study Day 30
  Clinical status assessed using a 7-category ordinal scale
Incidence of ADA | Study Day 30
  Defined as the precentage of subjects presenting anti-drug antibody

CONTACTS AND LOCATIONS:
Overall Officials: Bin Du, Principal Investigator — Peking Union Medical College Hospital; Huadong Zhu, Principal Investigator — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: No